CLINICAL TRIAL: NCT02055495
Title: Prospective Comparison of Subtalar Arthroereisis To Lateral Column Lengthening for Painful Flatfeet
Brief Title: Arthroereisis Versus Lateral Column Lengthening in the Treatment of Planovalgus Feet
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Bruce MacWilliams, Associate Professor, Director, Movement Analysis Laboratory, University of Utah
Other Study IDs: 40286
Record Dates: First submitted 2014-02-03; First posted 2014-02-05 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-08

CONDITIONS: Flatfeet
Keywords: Painful flatfeet; Planovagus feet; Subtalar arthroeresis; Lateral column lengthening; Kinematic motion analysis
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
There is no consensus on the surgical treatment of unremitting, painful flatfeet in children. Subtalar arthroereisis has gained notoriety although there is a paucity of literature on its biomechanical effects. The goal of the investigators was to compare a group treated with subtalar arthroereisis with another group undergoing lateral column calcaneal lengthening. The investigators hypothesis was that the results of arthroereisis would be equivalent to the more established method of calcaneal lengthening.

DETAILED DESCRIPTION:
The purpose of this prospective, non-randomized study was to evaluate two different surgical treatments for symptomatic planovalgus feet: lateral column lengthening osteotomy and subtalar arthroereisis. The goal of the investigators was to compare the outcomes of these two surgeries and determine whether both treatments resulted in clinical improvement. This was accomplished through the use of pre- and post-operative kinematics, pedobarography, radiographic measurements, and validated outcome measures. The investigators were particularly interested in analyzing the kinematic changes to quantify the changes in the foot mobility and alignment during ambulation, as it has not been previously studied to our knowledge. The investigators hypothesis was that both procedures would show significant improvement and be equivalent in their results.

A prospective trial was conducted. The investigators enrolled fifteen patients (mean age 12.8y, 24 feet) with painful, planovalgus feet refractory to conservative treatment. Seven patients (13 feet) were enrolled in the arthroereisis group, and eight patients (11 feet) were enrolled in the calcaneal lengthening group. Though not specifically excluded, none of the enrolled patients had an underlying neuromuscular diagnosis. Kinematic motion analysis was performed on each patient prior to surgery and at one year of follow-up. Pedobarometry studies, radiographs, and validated outcome questionnaires (Oxford Ankle-Foot Questionnaire for Children) were also performed to evaluate the outcomes of both groups.

ELIGIBILITY:
Inclusion Criteria:

* Planovalgus foot deformity
* Patient normally ambulates without use of assistive devices
* Patient is between the ages of 7 and 17 at the initial evaluation

Exclusion Criteria:

* Hip flexion contractures greater than 15 deg.
* Knee flexion contractures greater than 10 deg.
* Ankle dorsiflexion less than 0 deg. (plantarflexion contracture)
* Taking medication which effects motor control
* Inability to follow instructions to perform study

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patient ages ranged from 7 to 17 (mean 12.8y) at the time of surgery. Inclusion criteria were patients with planovalgus deformity, painful symptoms refractory to conservative treatment for at least 6 months, and independent ambulation without the use of assistive devices.
  A longitudinally study of two patient cohorts: 1) children with planovalgus foot deformity treated with arthroereisis (subtalar implant) and 2) children with planovalgus foot deformity treated by calcaneal (lateral column) lengthening.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2010-03; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Kinematics motion analysis | 1 year
  The change in hindfoot angle, degree of hindfoot mobility both pre- and postoperatively, degree of ankle motion both pre- and postoperatively, and amount of flexion occurring between the forefoot and hindfoot both pre- and postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce MacWilliams, Ph.D., Principal Investigator — University of Utah
Locations (1):
- Shriners Hospitals for Children, Salt Lake City, Utah, United States